CLINICAL TRIAL: NCT00967382
Title: TIPPS - Thrombophilia in Pregnancy Prophylaxis Study: A Multicentre, Multinational, Randomized Control Trial of Prophylaxis Low Molecular Weight Heparin (LMWH) in High-risk Thrombophilic Women.
Brief Title: TIPPS: Thrombophilia in Pregnancy Prophylaxis Study
Acronym: TIPPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1999210-01H; IND 72,350 (Other: Department of Health & Human Services, FDA); ISRCTN 87441504 (Registry Identifier: ISRCTN); CIHR 200602MCT-157533-RFA (Other Grant/Funding Number: Canadian Institutes of Health Research); Trial number 2004/244 (Other: Australian Government,Therapeutic Goods Administration); 2007-000284-21 (EudraCT Number)
Record Dates: First submitted 2009-05-29; First posted 2009-08-27 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Pregnancy; Thrombophilia; Pregnancy Complications
Keywords: Pregnancy; Thrombophilia; High-risk pregnancy; LMWH prophylaxis; Placenta mediated pregnancy complications
MeSH Terms: conditions — Thrombophilia; Pregnancy Complications | interventions — Dalteparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Subjects randomized to control will receive identical obstetrical care and follow-up, but not antenatal dalteparin.
  Within 24 hours of delivery, all subject's, regardless of randomization allocation will receive dalteparin sodium 5,000 IU s.c. daily for 6 weeks post-partum
- dalteparin sodium (Active Comparator): Subjects randomized to the treatment group will receive daily injections of dalteparin during the antenatal period. They will be taught how to self-administer sub-cutaneous injections of dalteparin 5000 IU once daily (o.d.) until gestational age 20, then twice daily (bid) until 37 weeks gestation or onset of labour.
  Within 24 hours of delivery, all subject's, regardless of randomization allocation will receive dalteparin sodium 5,000 IU s.c. daily for 6 weeks post-partum
  Interventions: Drug: dalteparin sodium

INTERVENTIONS:
Drug: dalteparin sodium — Subject's randomize to treatment arm will receive dalteparin sodium 5,000 IU s.c. daily starting on randomization day until 20 weeks gestational age then;
  dalteparin sodium 5,000 IU s.c. bid from 20 weeks to onset of labour or 37 weeks gestation (discontinued at the discretion of the investigator/obstetrician)
  Within 24 hours of delivery, all subject's, regardless of randomization allocation will receive dalteparin sodium 5,000 IU s.c. daily for 6 weeks post-partum
  Other Names: Fragmin
  Arms: dalteparin sodium

SUMMARY:
The TIPPS trial seeks to determine the safety and effectiveness of low-molecular-weight heparin (LMWH), an anticoagulant, in preventing placenta mediated pregnancy complications and venous thromboembolism (VTE) in women with thrombophilia. Thus, the principal research question is: can LMWH prevent thrombosis in the leg veins, pulmonary arteries and placental vessels, thereby reducing the risk of deep vein thrombosis, pulmonary embolism (PE), intrauterine growth restriction (IUGR), preeclampsia, miscarriage and stillbirth?

DETAILED DESCRIPTION:
TIPPS is a multicentre, multi-national open-label randomized controlled clinical trial. Two hundred and eighty-four thrombophilic women at risk for VTE or placenta mediated pregnancy complications will be recruited. Patients who require anticoagulant prophylaxis during this pregnancy (as judged by the local investigator) or have participated in TIPPS before will not be eligible for the trial.

The study consists of five periods: screening, randomization, antenatal follow-up, labour and delivery, and the post-partum follow-up.

Eligible and consenting patients will be assigned to one of two groups (treatment or control), stratified by gestational age at randomization: less than 8 weeks, 8 weeks +1 day to 12 weeks , 12 weeks +1 day to 19 weeks + 6 days.

Treatment Group - Subjects randomized to the treatment group will receive daily injections of dalteparin during the ante-natal period. They will be taught how to self-administer sub-cutaneous injections of dalteparin 5000 International units (IU) once daily (o.d.) until gestational week 20, then twice daily (bid) until 37 weeks gestation or onset of labour.

Control Group- Subjects randomized to control will receive identical obstetrical care and follow-up, but no ante-natal dalteparin.

Visit Schedule Subject will be evaluated for study eligibility and once the consent has been signed a baseline assessment will be completed. Randomization is done within 7 days of the baseline visit.

All patients will be seen in person for the first follow-up visit 7-9 days after randomization. Subsequent visits are based on the gestational age of the fetus and will be as follows:

* Monthly (+/- 1 week) from gestational week 8 to 28 -
* Every 2 weeks (+/- 1 week) from gestational week 28 to 34
* Every week from gestational week 35 until delivery.

The following visits are required in-person at day 7-9 and at gestational weeks 12, 20, 28, 32 and/or 36 and at 6 weeks post-partum to coincide with safety blood draws for hematology and biochemistry regardless of treatment allocation.

The remaining visits can be done in person or by phone calls: at gestational weeks 8, 16, 24, 30, 34, 35, 37, 38, 39 and 40. If available, results for hematology and biochemistry done at gestational age 8, 16, 24 and 40 will be recorded.

At each visit, weight and blood pressure measurements will be recorded and all subjects will be monitored for study progress, study outcomes, adverse events (AEs), and concomitant medications. Subjects randomized to receive dalteparin will have their compliance assessed through the monthly visits. Subjects will be required to complete the patient injection diary and will be asked to bring it with them at all in-person-visits. The diary will be collected at the completion of study participation.

Labour and delivery: outcomes and AEs will be assessed through a review of subjects' medical records. If available, results from blood drawn for hematology and biochemistry will be recorded. Data pertaining to the labour and delivery, as well as foetal weight and health at birth, will be documented. For those subjects randomized to receive dalteparin, the date and time of the last injection will be noted.

During the six-week postpartum period, all subjects will receive dalteparin 5,000 IU o.d. for VTE prophylaxis. Subjects randomized to control will be taught to self-administer the subcutaneous injections prior to starting their postpartum injections. Subjects will be asked to complete the patient injection diary and to return it at the final visit. The final study visit occurs at 6 weeks post-partum (+/- 1week) or at early termination; at this visit study progress, study outcomes, adverse events, results from blood drawn for hematology and biochemistry and compliance with study drug will be documented.

ELIGIBILITY:
Inclusion Criteria:

One or more of the following:

* Previous preeclampsia
* Previous unexplained intra-uterine growth restriction
* Previous recurrent miscarriage:

  * three(3) or more unexplained miscarriage at less than 10 weeks gestation;
  * two (2) or more unexplained fetal loss between 10 and 16 weeks gestation;
  * one (1) or more unexplained fetal loss at or greater than 16 weeks gestation
* Previous abruptio placenta
* Previous personal history of VTE:

  * Previous documented secondary proximal VTE,
  * Previous documented calf-vein thrombosis (idiopathic or secondary),
  * Previous superficial phlebitis
* First degree relative with symptomatic thrombophilia
* Pregnancy - > 4weeks gestation and < 20 weeks gestation
* Thrombophilia:
* Two abnormal tests, and no normal tests

  * 3.1 Protein S
  * 3.2 Protein C
  * 3.3 Antithrombin
* Two positive tests

  * 3.4 Anticardiolipin immunoglobulin M (IgM) (>30 U/ml)
  * 3.5 Anticardiolipin immunoglobulin G (IgG) (>30 U/ml)
  * 3.6 Anti-b2 glycoprotein IgG (>20 U/ml)
  * 3.7 Anti-b2 glycoprotein IgM (>20 U/ml)
  * 3.8 Lupus anticoagulant
* One positive test

  * 3.9 Factor V Leiden (heterozygous or homozygous)
  * 3.10Prothrombin gene defect (heterozygous or homozygous)

Exclusion Criteria:

* Less than 4 weeks gestation or greater than 20 weeks gestation
* No confirmed thrombophilia
* Contraindication to heparin therapy

  * History of heparin induced thrombocytopenia
  * Platelet count less than 100,000 109/L
  * History of osteoporosis or steroid use
  * Actively bleeding
  * Documented peptic ulcer within 6 weeks
  * Heparin, bisulfite or fish allergy
  * Severe hypertension (Systolic Blood Pressure >200mmhg and/or Diastolic Blood Pressure >120mmHg)
  * Serum creatinine greater than 80 umol/L (1.3mg/dl) and an abnormal 24 hour urine creatine clearance (<30ml/min)
  * Severe hepatic failure (INR >1.8)
* Geographic inaccessibility
* Need for anticoagulants, discretion of the investigator such as but not limited to:

  * Recurrent fetal loss and phospholipid antibody syndrome
  * Prior idiopathic proximal VTE:
  * History of idiopathic deep venous thrombosis (DVT) or pulmonary embolism (PE) treated with anticoagulants (> 1 month of heparin or warfarin) or inferior vena cava (IVC) interruption;
  * Idiopathic is a VTE occurring outside all of the following periods: antepartum, postpartum, oral contraceptive use, surgery, immobilization, cast, and malignancy
  * Mechanical heart valve
* Legal lower age limitations (country specific)
* Prior participation in TIPPS
* Unable/unwilling to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2000-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to identify if LMWH prophylaxis in thrombophilic pregnant women results in a greater than 33% relative risk reduction in the composite outcome measure (VTE, pre-eclampsia, IUGR and fetal loss) | 6 weeks post-partum

SECONDARY OUTCOMES:
Identify if prophylactic LMWH will reduce rates of pregnancy induced hypertension (PIH), preterm labor and abruptio placenta in pregnant thrombophilic women compared to control | 6 weeks post-partum
Determine the safety of LMWH use in pregnancy (Specifically rates of bleeding, thrombocytopenia and fractures) | 6 weeks post-partum
Identify whether prolonged use of LMWH in pregnancy results in decreased bone mineral density (BMD) compared to control | 6 weeks post-partum

CONTACTS AND LOCATIONS:
Overall Officials: Marc A Rodger, MD, Principal Investigator — Ottawa Hospital Research Institute, Ottawa, Canada; William Hague, MD, Principal Investigator — Women's and Children's Hospital, Adelaide, Australia
Locations (12):
- United States (2):
  - Saint Louis University, St Louis, Missouri
  - University of Utah Health Sciences Centre, Salt Lake City, Utah
- Canada (10):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - The Ottawa Hospital, Civic Campus, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Women's College Health Sciences Centre, Toronto, Ontario
  - SMBD Jewish General Hospital, Montreal, Quebec
  - St Mary's Hospital Centre, Montreal, Quebec
  - CHA, Hopital Enfant Jesus, Québec, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Middleton P, Shepherd E, Gomersall JC. Venous thromboembolism prophylaxis for women at risk during pregnancy and the early postnatal period. Cochrane Database Syst Rev. 2021 Mar 29;3(3):CD001689. doi: 10.1002/14651858.CD001689.pub4. PMID 33779986
- [Derived] Rodger MA, Hague WM, Kingdom J, Kahn SR, Karovitch A, Sermer M, Clement AM, Coat S, Chan WS, Said J, Rey E, Robinson S, Khurana R, Demers C, Kovacs MJ, Solymoss S, Hinshaw K, Dwyer J, Smith G, McDonald S, Newstead-Angel J, McLeod A, Khandelwal M, Silver RM, Le Gal G, Greer IA, Keely E, Rosene-Montella K, Walker M, Wells PS; TIPPS Investigators. Antepartum dalteparin versus no antepartum dalteparin for the prevention of pregnancy complications in pregnant women with thrombophilia (TIPPS): a multinational open-label randomised trial. Lancet. 2014 Nov 8;384(9955):1673-83. doi: 10.1016/S0140-6736(14)60793-5. Epub 2014 Jul 24. PMID 25066248
- [Derived] Bennett SA, Bagot CN, Arya R. Pregnancy loss and thrombophilia: the elusive link. Br J Haematol. 2012 Jun;157(5):529-42. doi: 10.1111/j.1365-2141.2012.09112.x. Epub 2012 Mar 26. PMID 22449204
- See also: The Ottawa Hospital Research Institute is the sponsor for TIPPS. This site provides information about the lead institution and provides a link the to coordinating centre located within the thrombosis program. — http://www.ohri.ca/home.asp
- See also: Site of the Canadian Institutes of Health Research - information regarding the terms of reference related to the TIPPS grant can be found herein. — http://cihr-irsc.gc.ca